CLINICAL TRIAL: NCT01363154
Title: Prevention of Photoparoxysmal Abnormalities Through Patterned Auditory Stimulation
Brief Title: Prevention of Photoparoxysmal Abnormalities by Mozart K448
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Robert P. Turner, Assoc Prof Neurosciences, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7683
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Photoparoxysmal Abnormalities; Epilepsy; Seizures
Keywords: Children's Health; Pediatrics; Epilepsy; Photoparoxysmal; Photosensitive; Music; Mozart; K-448
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mozart K448 (Active Comparator): Treatment: music exposure to Mozart K448
  Interventions: Other: Mozart K448
- Beethoven's Für Elise (Placebo Comparator): Placebo: music exposure to Beethoven's Für Elise for piano
  Interventions: Other: Beethoven's Für Elise; Other: No music exposure
- No music exposure (No Intervention): Control: no music exposure

INTERVENTIONS:
Other: Mozart K448 — Subjects will receive auditory stimulation by exposure to Mozart's Sonata for Two Pianos in D Major, K448.
  Other Names: Mozart's Sonata for Two Pianos in D Major, K448
  Arms: Mozart K448
Other: Beethoven's Für Elise — Subjects will receive auditory stimulation by exposure to Beethoven's Für Elise.
  Arms: Beethoven's Für Elise
Other: No music exposure — Subject's will not receive an intervention and will therefore, not receive auditory stimulation and/or exposure to music.
  Other Names: Control: No music exposure.
  Arms: Beethoven's Für Elise

SUMMARY:
The purpose of this clinical trial is to examine the effect of non-invasive cortical activation by specific patterned auditory stimulation (Mozart K448- Piano Sonata for Two Hands in D Major), in altering or eliminating photoparoxysmal abnormalities. Recent work has indicated that such evoked activity (i.e. by specific music) can result in significant reductions, or even complete termination of epileptiform activity and/or seizures across a broad range of individuals with epilepsy. A hypothesis is generated that specific music activation would beneficially effect photoparoxysmal based epileptiform abnormalities.

DETAILED DESCRIPTION:
Non-pharmacologic, non-surgical treatments for seizures and epilepsy are of increasing importance, given the potential side effects as well as lack of complete seizure control with such treatments. Based on previous studies demonstrating an anti-convulsant and anti-epileptiform effect achieved in subjects by music exposure, it is proposed that specific musical stimuli may causally result in widely distributed cortical activation in such a fashion as to effectively prevent or terminate epileptiform abnormalities in subjects with photosensitive epilepsy. We will investigate the effect of specific musical stimulation (Mozart K448) to reduce or prevent photoparoxysmal abnormalities in subjects.

Primary outcome will be evaluated in 3 groups, assessing alteration/cessation of photic-induced abnormalities during:

1. Treatment: music exposure to Mozart K448, vs.
2. Placebo: music exposure to Beethoven's Für Elise for piano, vs.
3. Control: no music exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-17 years, inclusive
* Female or male with photoparoxysmal epilepsy clinical history, and at least one seizure, as defined by the International League Against Epilepsy (International Classification of Epilepsies and Epileptic Syndromes; Commission on Classification and Terminology of the International League Against Epilepsy 1989)
* Abnormal EEG consistent with features of photoparoxysmal epilepsy: occipital based epileptiform abnormalities with otherwise normal background interictal EEG;
* On < or equal to 2 anti-seizure medications [range 0-2 AEDs]

Exclusion Criteria:

* History of a generalized convulsion provoked by photic stimulation;
* Inability to complete and/or comply with study protocol

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Decreased duration (>25%) of photoparoxysmal response(s) during exposure to K-448 | Each participant will have a single one hour EEG for data aquistition.
  Each participant will have a single one hour EEG for data aquistition. The recorded EEG data will be analyzed to determine significant causal reductions or prevention of photoparoxysmal responses resulting from the auditory stimulation, along with determining all induced patterns of cortical activation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Turner, MD, MSCR, Principal Investigator — Medical University of South Carolina; Mark Bodner, MD, Principal Investigator — MIND Institute; Lee Anne Tetrick, BS, Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Banerjee PN, Filippi D, Allen Hauser W. The descriptive epidemiology of epilepsy-a review. Epilepsy Res. 2009 Jul;85(1):31-45. doi: 10.1016/j.eplepsyres.2009.03.003. Epub 2009 Apr 15. PMID 19369037
- [Background] Bodner M, Muftuler LT, Nalcioglu O, Shaw GL. FMRI study relevant to the Mozart effect: brain areas involved in spatial-temporal reasoning. Neurol Res. 2001 Oct;23(7):683-90. doi: 10.1179/016164101101199108. PMID 11680506
- [Background] Davis R, Emmonds SE. Cerebellar stimulation for seizure control: 17-year study. Stereotact Funct Neurosurg. 1992;58(1-4):200-8. doi: 10.1159/000098996. PMID 1439341
- [Background] Engel J Jr; International League Against Epilepsy (ILAE). A proposed diagnostic scheme for people with epileptic seizures and with epilepsy: report of the ILAE Task Force on Classification and Terminology. Epilepsia. 2001 Jun;42(6):796-803. doi: 10.1046/j.1528-1157.2001.10401.x. No abstract available. PMID 11422340
- [Background] Fisher RS, Uematsu S, Krauss GL, Cysyk BJ, McPherson R, Lesser RP, Gordon B, Schwerdt P, Rise M. Placebo-controlled pilot study of centromedian thalamic stimulation in treatment of intractable seizures. Epilepsia. 1992 Sep-Oct;33(5):841-51. doi: 10.1111/j.1528-1157.1992.tb02192.x. PMID 1396427
- [Background] Fisher RS, Harding G, Erba G, Barkley GL, Wilkins A; Epilepsy Foundation of America Working Group. Photic- and pattern-induced seizures: a review for the Epilepsy Foundation of America Working Group. Epilepsia. 2005 Sep;46(9):1426-41. doi: 10.1111/j.1528-1167.2005.31405.x. PMID 16146439
- [Background] Hughes JR, Daaboul Y, Fino JJ, Shaw GL. The "Mozart effect" on epileptiform activity. Clin Electroencephalogr. 1998 Jul;29(3):109-19. doi: 10.1177/155005949802900301. PMID 9660010
- [Background] Hughes JR, Fino JJ, Melyn MA. Is there a chronic change of the "Mozart effect" on epileptiform activity? A case study. Clin Electroencephalogr. 1999 Apr;30(2):44-5. doi: 10.1177/155005949903000204. PMID 10358782
- [Background] Hughes JR. The Mozart Effect. Epilepsy Behav. 2001 Oct;2(5):396-417. doi: 10.1006/ebeh.2001.0250. PMID 12609277
- [Background] Hughes JR. The Mozart Effect: Additional Data. Epilepsy Behav. 2002 Apr;3(2):182-184. doi: 10.1006/ebeh.2002.0329. PMID 12609420
- [Background] Jacobs MP, Fischbach GD, Davis MR, Dichter MA, Dingledine R, Lowenstein DH, Morrell MJ, Noebels JL, Rogawski MA, Spencer SS, Theodore WH. Future directions for epilepsy research. Neurology. 2001 Nov 13;57(9):1536-42. doi: 10.1212/wnl.57.9.1536. PMID 11706087
- [Background] Lahiri N, Duncan JS. The Mozart effect: encore. Epilepsy Behav. 2007 Aug;11(1):152-3. doi: 10.1016/j.yebeh.2007.04.017. Epub 2007 Jun 29. PMID 17602882
- [Background] Macdonell RA, Curatolo JM, Berkovic SF. Transcranial magnetic stimulation and epilepsy. J Clin Neurophysiol. 2002 Aug;19(4):294-306. doi: 10.1097/00004691-200208000-00004. PMID 12436086
- [Background] Kasteleijn-Nolst Trenite DG, Binnie CD, Harding GF, Wilkins A. Photic stimulation: standardization of screening methods. Epilepsia. 1999;40 Suppl 4:75-9. doi: 10.1111/j.1528-1157.1999.tb00911.x. PMID 10487178
- [Background] Kasteleijn-Nolst Trenite DG, van der Beld G, Heynderickx I, Groen P. Visual stimuli in daily life. Epilepsia. 2004;45 Suppl 1:2-6. doi: 10.1111/j.0013-9580.2004.451004.x. PMID 14706037
- [Background] Sarnthein J, vonStein A, Rappelsberger P, Petsche H, Rauscher FH, Shaw GL. Persistent patterns of brain activity: an EEG coherence study of the positive effect of music on spatial-temporal reasoning. Neurol Res. 1997 Apr;19(2):107-16. doi: 10.1080/01616412.1997.11740782. PMID 9175137
- [Background] Thornton-Wells TA, Cannistraci CJ, Anderson AW, Kim CY, Eapen M, Gore JC, Blake R, Dykens EM. Auditory attraction: activation of visual cortex by music and sound in Williams syndrome. Am J Intellect Dev Disabil. 2010 Mar;115(2):172-89. doi: 10.1352/1944-7588-115.172. PMID 20440382
- [Background] Turner RP. The acute effect of music on interictal epileptiform discharges. Epilepsy Behav. 2004 Oct;5(5):662-8. doi: 10.1016/j.yebeh.2004.07.003. PMID 15380117
- [Background] Van Buren JM, Wood JH, Oakley J, Hambrecht F. Preliminary evaluation of cerebellar stimulation by double-blind stimulation and biological criteria in the treatment of epilepsy. J Neurosurg. 1978 Mar;48(3):407-16. doi: 10.3171/jns.1978.48.3.0407. No abstract available. PMID 344840
- [Background] Verduzco-Flores S, Ermentrout B, Bodner M. From working memory to epilepsy: dynamics of facilitation and inhibition in a cortical network. Chaos. 2009 Mar;19(1):015115. doi: 10.1063/1.3080663. PMID 19335019
- [Background] Bodner M, Turner RP, Bowers C, Norment C (2009) Patterned auditory stimulus reduces seizure frequency in neurologically-impaired individuals. (submitted May 2010 to Epilepsia for publication)
- [Background] CURE: Citizens United for Research in Epilepsy. Web. 04 Oct. 2010. <http://www.cureepilepsy.org/home.asp>.
- [Background] Epilepsy Foundation of America. Web. 04 Oct. 2010. <https://efa.org/>.
- [Background] Franaszczuk PJ, Kudela P, Bergey GK. External excitatory stimuli can terminate bursting in neural network models. Epilepsy Res. 2003 Feb;53(1-2):65-80. doi: 10.1016/s0920-1211(02)00248-6. PMID 12576169
- [Background] Harding GF, Jeavons PM. Photosensitive Epilepsy. MacKeith Press, London, 1994.
- [Background] Temkin O. The falling sickness: A history of epilepsy from the Greeks to the beginnings of modern neurology. Baltimore: Johns Hopkins University Press, 1971.
- [Background] Turner RP, Bodner M, Wang L, Norment C, Bowers C, Zhou Y. The anti-epileptiform effect of acute auditory stimulation on Rolandic spikes: EEG spectral analysis and coherence in patients with Rolandic epilepsy. (2010 in preparation)
- [Background] ILAE: International League Against Epilepsy. Web. 02 Oct. 2010. <http://www.ilae-epilepsy.org/>.
- [Background] Zifkin BG and Andermann F. Visual Sensitive Epilepsies. International League Against Epilepsy. 28 Feb. 2005. Web. 04 Oct. 2010. <http://www.ilae-epilepsy.org/>.